CLINICAL TRIAL: NCT03040180
Title: Endoscopic Assisted Electrochemotherapy in Addition to Neoadjuvant Treatment of Locally Advanced Rectal Cancer: a Randomized Clinical Phase II Trial
Brief Title: Endoscopic Assisted Electrochemotherapy in Addition to Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Acronym: nECT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-32-2016
Record Dates: First submitted 2017-01-25; First posted 2017-02-02 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Locally Advanced Rectal Cancer; Electrochemotherapy; Neoadjuvant Therapy; Down Staging
Keywords: Neoplasms; Neoplasms, primary; Cancer; Colorectal cancer; rectal cancer; rectal cancer, locally advanced; Electrochemotherapy; Electroporation; Neoadjuvant therapy; Antineoplastic, antibodies; Bleomycin; Pathologic processes; Neoplastic processes
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Rectal Neoplasms; Pathologic Processes; Neoplastic Processes | interventions — Electrochemotherapy; Bleomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrochemotherapy with bleomycin (Experimental): Systemic injection of bleomycin followed by electroporation of the primary tumor. Bleomycin administration: 15.000 IU/m2 BSA.
  BSA by Du Bois formula.
  Interventions: Drug: Electrochemotherapy with bleomycin; Device: EndoVE
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Drug: Electrochemotherapy with bleomycin — Systemic injection, once only treatment
  Other Names: ATC code L01DC01; EV substance code SUB00844MIG
  Arms: Electrochemotherapy with bleomycin
Device: EndoVE — Electroporation using an endoscopic electroporation device
  Other Names: Endoscopic electroporation
  Arms: Electrochemotherapy with bleomycin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of neoadjuvant electrochemotherapy on locally advanced rectal cancer (UICC II-III) in an intended curative clinical setting, using an endoscopic electroporation device (EndoVE).

DETAILED DESCRIPTION:
Electroporation of cancer cells allows for a greater concentration of chemotherapy drugs to enter the tumor cells. The uptake of the chemotherapeutic drug is aided through the application of short electric pulses to the tumor mass (referred to as - Electrochemotherapy or ECT). The pulses make the tumor cells more porous which allows the drug easier access into the cancer cells, whereas other tissues and organs in the body remain relatively poor at absorbing the drug, thereby reducing the potential side effects on healthy tissues. Procedures with electrochemotherapy have previously been applied to human patients in other countries of the EU, the US and Japan.

The drug concentration used is significantly reduced due to the more targeted absorption by the tumor and this significantly reduces side effects normally associated with chemotherapy.

A large number of preclinical and clinical Phase I and I/II studies have demonstrated the efficiency and safety of ECT. These studies have included patients with melanoma, head and neck squamous cell carcinoma, merkel cell carcinomas, basal cell carcinoma and adenocarcinoma nodules.

An endoscopic system (EndoVE ) for delivering the electric pulses to gastrointestinal tumors has recently been developed. The treatment procedure is similar to standard endoscopic colorectal examination (therapeutic colonoscopy) with the added element of an intravenous injection of bleomycin followed by the delivery of electric pulses (each one less than 1msec in duration). The pulses are endoscopically delivered directly to the tumor mass. The entire procedure is minimally invasive and completely ambulatory. A successful treatment will cause the tumor to shrink in size in the weeks following the procedure.

The objective of this study is to investigate the efficacy and safety of this approach in downsizing locally advanced rectal tumors prior to intended curative surgery.

Time frame:

1. All patients will be treated with standard neoadjuvant chemoradiation therapy prior to enrollment in this trial.
2. Alle patients will have PET/MRI scans performed twice to evaluate treatment response (before and after ECT)
3. ECT treatment will be performed 4 weeks prior to surgery outlined by MDT.
4. Alle patients will be followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be mentally capable of understanding the information given.
2. Patients must give written informed consent.
3. Men or women aged at least 18 years.
4. Histologically verified rectal tumor (adenocarcinoma)
5. Case reviewed by MDT (surgery, radiology, oncology). Case considered curable with neoadjuvant therapy followed by surgical excision (UICC stadium II-III).
6. ASA class I-III (Classification of the American Society of Anesthesiology)

Exclusion Criteria:

1. Coagulation disorders
2. Highly inflamed gastrointestinal tissue which is ulcerated and bleeding
3. Patients with ICD or pacemaker units.
4. Patients with epilepsy.
5. Pregnancy or lactation/breastfeeding.
6. Patients with known Hepatitis B/C or HIV infection.
7. Patients who have undergone treatment with bevacizumab within 4 weeks prior to enrolment in this trial.
8. Patients with concomitant use of phenytoin.
9. Patients with concomitant use of clozapine.
10. Concurrent treatment with an investigational medicinal product.
11. Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study recruitments.
12. Patients with contraindications for PET/MRI scan:
13. Advanced tumor stage, UICC stage IV.
14. Acute pulmonary infection.
15. Medical history of severe pulmonary disease.
16. Previous allergic reactions to bleomycin.
17. Previous cumulative dose of bleomycin exceeding 250.000 IU/m2.
18. Pre-existing renal dysfunction. Creatinine clearance < 40 ml/min.
19. Platelet count ≤50 mia/l.
20. Prothrombin time ≥ 40 sec
21. Patients registered in the Danish Tissue Register (Vaevsanvendelsesregistret)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Histopathologic tumor regression following electrochemotherapy | 4 weeks
  Number of participants with histopathologic tumor regression following elctrochemotherapy as assesed by histopathological evaluation of Tumor Regression Grade (Mandard Classification, TRG 1-5)

SECONDARY OUTCOMES:
Treatment safety of electrochemotherapy | 4 months
  Number of participants with treatment-related adverse events as assesed by CTCAE version 4.0
Treatment safety of surgery following electrochemotherapy | 4 weeks
  Number of participants with compromized surgery following electrochemotherapy assesed by R1 resection rate, CRM involvement, non-mesorectal resection plane, and post operative complications according to Clavien-Dindo Classification
Tumor regression according to Hybrid PET/MRI following electrochemotherapy | 4 weeks
  Tumor regression as assesed by tumor stage (T-stage)
Tumor Immunologic response following electrochemotherapy | 4 weeks
  Tumor immunologic infiltration as assesed by the Immunoscore through immunohistochemical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Professor, Principal Investigator — Department of Surgery, Zealand University Hospital; Julie Gehl, MD, DMSc, Principal Investigator — Department of oncology, herlev Hospital
Locations (2):
- Denmark (2):
  - Department of Oncology, Herlev, Capitol Region
  - Department of Surgery, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided
Undecided